CLINICAL TRIAL: NCT04135339
Title: Efficacy of Exercise on Post Needling Soreness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Nicola Sante Diciolla, Physiotherapist, Master of Sciences, Associate Researcher, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEI/HU/2019/27
Record Dates: First submitted 2019-09-22; First posted 2019-10-22 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Post Needling Soreness; Myofascial Pain; Myofascial Pain Syndrome; Myofascial Trigger Point Pain
Keywords: pain; trigger points; physical therapy; dry needling; therapeutic exercise
MeSH Terms: conditions — Myofascial Pain Syndromes; Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A. Eccentric exercise. (Experimental): 15 subjects with a latent myofascial trigger point in the medial gastrocnemius muscle.
  Interventions: Other: Eccentric exercise
- Group B. Concentric exercise. (Experimental): 15 subjects with a latent myofascial trigger point in the medial gastrocnemius muscle.
  Interventions: Other: Concentric exercise.
- Group C. Isometric exercise. (Experimental): 15 subjects with a latent myofascial trigger point in the medial gastrocnemius muscle.
  Interventions: Other: Isometric exercise.
- Group D. Control. (No Intervention): 15 subjects with a latent myofascial trigger point in the medial gastrocnemius muscle.

INTERVENTIONS:
Other: Eccentric exercise — The exercise session will consist of 3 sets of 15 reps, 3´´ per rep, with 30'' rest between sets, of the previous treated gastrocnemius muscle (by DN). Each rep will be a pure eccentric contraction.
  Arms: Group A. Eccentric exercise.
Other: Concentric exercise. — The exercise session will consist of 3 sets of 15 reps, 3´´ per rep, with 30'' rest between sets, of the previous treated gastrocnemius muscle (by DN). Each rep will be a pure concentric contraction.
  Arms: Group B. Concentric exercise.
Other: Isometric exercise. — The exercise session will consist of 3 sets of 15 reps, 3´´ per rep, with 30'' rest between sets, of the previous treated gastrocnemius muscle (by DN). Each rep will be a pure isometric contraction.
  Arms: Group C. Isometric exercise.

SUMMARY:
Introduction. The myofascial trigger point (MTrP) is a clinical entity related to different clinical pictures of pain. Dry needling (DN) would be the most appropriate therapeutic option for its treatment, although it has mild-moderate adverse effects, such as post-needling soreness (PNS). The exercise could be a strategy for its management, but no recommendations on the most effective mode have been found.

Objectives

1. To determine the effectiveness of the exercise, differentiated according to the dominant mode (concentric, eccentric, isometric), in order to reduce the PNS of latent MTrPs.
2. To analyse the variables that, a priori, can influence the evolution of pain.

Methods. Study design .A randomized clinical trial. Scenario Private or home-based consultation in Global Physiotherapy, Madrid, Spain.

Participants. Voluntaries, with no symptoms in the triceps surae muscle,>18 years old, who present at least one latent MTrP in medial gastrocnemius. Subjects with: other pathologies of lower limbs, active MTrP in the medial gastrocnemius muscle, contraindications to DN, prior application of DN and/or other therapies in MTrPs during the three months previous to the study (in gastrocnemius muscles) will be excluded.

Intervention After DN of the medial gastrocnemius muscle, participants will be randomly allocated to four groups (three experimental groups and one control). In the experimental groups, subjects will be instructed to perform exercise protocols, differentiated according to the dominant contraction (concentric, eccentric, isometric) in muscle the gastrocnemius previously treated.

Outcome measures. Pain intensity, by analog visual scale (VAS). Pressure pain threshold (PPT), by analog algometer. Demographics and anthropometrics.

Protocol. Before and immediately after DN, the PPT will be evaluated in the latent MTrP. Pain intensity will also be assessed using VAS at two times: the first referred to pain during DN and the other referred to PNS two minutes after DN. The subjects will then be randomly divided into: a control group without any intervention after DN, and three experimental groups with different exercise protocols (differentiated by the dominant contraction: 3 sets x 15 reps, 3s each contraction, 30s of rest between sets) . The pain intensity will be recorded again by VAS, after the exercise session and at 6h, 12h, 24h, 48h, 72h after DN. PPT will also be assessed 2min after DN, after the exercise session and at 24h, and 48h after DN.

DETAILED DESCRIPTION:
Introduction. The myofascial trigger point (MTrP) is a clinical entity related to different clinical pictures of pain. Dry needling (DN) would be the most appropriate therapeutic option for its treatment, although it has mild-moderate adverse effects, such as post-needling soreness (PNS). The exercise could be a strategy for its management, but no recommendations on the most effective mode have been found.

Objectives

1. To determine the effectiveness of the exercise, differentiated according to the dominant mode (concentric, eccentric, isometric), in order to reduce the PNS of latent MTrPs.
2. To analyse the variables that, a priori, can influence the evolution of pain.

Methods Study design A randomized clinical trial. Scenario Private or home-based consultation in Global Physiotherapy, Madrid, Spain.

Participants. Voluntaries, with no symptoms in the triceps surae muscle,>18 years old, who present at least one latent MTrP in medial gastrocnemius. Subjects with: other pathologies of lower limbs, active MTrP in the medial gastrocnemius muscle, contraindications to DN, prior application of DN and/or other therapies in MTrPs during the three months previous to the study (in gastrocnemius muscles) will be excluded.

Intervention After DN of the medial gastrocnemius muscle, participants will be randomly allocated to four groups (three experimental groups and one control). In the experimental groups, subjects will be instructed to perform exercise protocols, differentiated according to the dominant contraction (concentric, eccentric, isometric) in muscle the gastrocnemius previously treated.

Outcome measures. Pain intensity, by analog visual scale (VAS). Pressure pain threshold (PPT), by analog algometer. Demographics and anthropometrics.

Protocol. Before and immediately after DN, the PPT will be evaluated in the latent MTrP. Pain intensity will also be assessed using VAS at two times: the first referred to pain during DN and the other referred to PNS two minutes after DN. The subjects will then be randomly divided into: a control group without any intervention after DN, and three experimental groups with different exercise protocols (differentiated by the dominant contraction: 3 sets x 15 reps, 3s each contraction, 30s of rest between sets) . The pain intensity will be recorded again by VAS, after the exercise session and at 6h, 12h, 24h, 48h, 72h after DN. PPT will also be assessed 2min after DN, after the exercise session and at 24h, and 48h after DN.

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least one latent myofascial trigger point (MTrP) in the medial gastrocnemius muscle.

Exclusion Criteria:

* Other lower limb pathologies which no permit the application of the interventions (e.g. lower limb fractures; sprain in acute phase; etc).
* Active MTrPs in the medial gastrocnemius muscle (related to tendinopathies, plantar fascitis).
* Fibromyalgia.
* Osteosynthesis materials.
* Pregnancy.
* Fear of needles.
* Previous application of dry needling (in gastrocnemius muscles).
* Other treatments of MTrPs during the three months previous to the study (in gastrocnemius muscles).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Change of post needling soreness. | 2 minutes after dry needling, just after exercise session (not for control group), 6 hours after exercise session, 12 hours after exercise session, 24 hours after dry exercise session, 48 hours after exercise session, 72 hours after exercise session.
  Visual analog scale (VAS) of 100 mm: 0 mm indicates absence of post needling soreness and 100 mm indicates maximum post needling soreness intensity

SECONDARY OUTCOMES:
Change of pressure pain threshold after dry needling. | 2 minutes after dry needling, just after exercise session (not for control group), 24 hours after exercise session, 48 hours after exercise session.
  Analog algometer (kilograms/squared centimeters -kg/cm2-).

OTHER OUTCOMES:
Pain intensity during dry needling | Before exercise session (i.e. during dry needling).
  Visual analog scale (VAS) of 100 mm: 0 mm indicates absence of pain and 100 mm indicates maximum pain intensity.
Pressure pain threshold before dry needling | Before intervention (i.e. dry needling and exercise session).
  Analog algometer (kilograms/squared centimeters -kg/cm2-).
Demographic data. | First assessment before intervention (i.e. dry needling and exercise session).
  Age (years).
Demographic data. | First assessment before intervention (i.e. dry needling and exercise session).
  Gender (male/female).
Anthropometric data. | First assessment before intervention (i.e. dry needling and exercise session).
  Height (meters -m-).
Anthropometric data. | First assessment before intervention (i.e. dry needling and exercise session).
  Weight (kilograms-kg-).

CONTACTS AND LOCATIONS:
Overall Officials: María Torres Lacomba, PT, PhD, Study Director — University of Alcalá, Madrid, Spain.
Locations (1):
- Nicola Sante Diciolla, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be available to those researchers who are interested in researching about the exercise effects on post needling soreness mailing with one of the members of the research group.
Supporting Information: Study Protocol, SAP
Time Frame: 1 year
Access Criteria: * Research interest in effects of exercise on post needling soreness.
  * Ethical Committee approval.